CLINICAL TRIAL: NCT06148779
Title: Can Digitally Delivered First-line Osteoarthritis Treatment Improve Equal Access to Care in Urban and Rural Areas of Sweden
Brief Title: Can Digitally Delivered First-line Osteoarthritis Treatment Improve Equal Access to Care
Acronym: Access
Status: Recruiting | Type: Observational
Sponsor: Joint Academy (Industry)
Collaborators: Lund University (Other); The Swedish Osteoarthritis Registry (Unknown)
Responsible Party: Sponsor
Other Study IDs: Access to care OA
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Health Services Accessibility; First-line Treatment; Osteoarthritis
Keywords: Osteoarthritis; Digitally delivered; Tele-health; Physiotherapy; Access to care; Exercise
MeSH Terms: conditions — Osteoarthritis; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Joint Academy
  Interventions: Behavioral: Digitally delivered first-line treatment for osteoarthritis
- BOA
  Interventions: Behavioral: Face-to-face first-line treatment for osteoarthritis

INTERVENTIONS:
Behavioral: Digitally delivered first-line treatment for osteoarthritis — Digitally delivered first-line for osteoarthritis through the caregiver Joint Academy.
  Groups: Joint Academy
Behavioral: Face-to-face first-line treatment for osteoarthritis — First-line for osteoarthritis delivered at a primary care clinic face-to-face with reported data to the BOA registry.
  Groups: BOA

SUMMARY:
To improve chronically ill patients' health and quality of life, long-standing and continuous treatment is needed at an acceptable cost. The purpose of this study was to compare utilization of digital versus face-to-face delivered osteoarthritis (OA) treatment in the 21 different county councils of Sweden that are responsible for providing healthcare to the residents.

DETAILED DESCRIPTION:
Since 2008 Sweden has had a structured first-line face-to-face knee and hip osteoarthritis (OA) treatment program, Better management of patients with OsteoArthritis (BOA). However, records show that this face-to-face program is underutilized and reaches only a minority of those that would benefit from it.

The first-line OA management program has been transformed into a digital version, Joint Academy® (JA), to facilitate implementation, scaling, increased accessibility, and improved patient adherence. The mobile application (app) consists of video instructions distributed daily with individualized exercises for participants with knee or hip OA, as well as educational information on OA symptoms and self-management based on current international guidelines for the management of OA. Each participant is assigned to a physical therapist available through asynchronous chat and telephone who supervises the participant throughout the whole program.

To improve chronically ill patients' health and quality of life, long-standing and continuous treatment is needed at an acceptable cost. Recent evidence suggests that JA costs 25% compared to the BOA program for three months of treatment. Providing patients with equal access to care necessitates availability in urban and rural areas alike. This can potentially be achieved by digital delivery, but it is yet unknown if digital delivery of first-line OA treatment, compared with face-to-face, improves equal access to care. The purpose of this study was to compare utilization of digital and face-to-face delivered OA treatment in the 21 different county councils of Sweden that are responsible for providing healthcare to the residents.

Method Registered patient participation in the BOA program during 2021-2023 will be retrieved from the BOA Register. The BOA registry. Data from digital program participation was retrieved from the JA database. To be included, a patient need to have registered for the first visit in the BOA registry or have enrolled in the program by answering the first questionnaire in the JA registry.

Population density per county and county size were retrieved from Statistics Sweden. Results were calculated and presented as users per 100 000 residents. Mean and median values as well as standard deviations were calculated separately for registered participants/100 000 for BOA and JA programs, and for regions with more (n=12) or less (n=8) than 20 residents per km2.

Please not that the BOA registry was in January 2023 renamed to The Swedish Osteoarthritis Registry.

ELIGIBILITY:
* Patients in the Joint Academy database that had participated in the Joint Academy treatment program for OA and given their informed consent to participate in research.

Inclusion criteria for the treatment program:

* Radiographic and or clinical diagnosis of hip or knee OA from a physical therapist or physician (95% of all patients in previously published studies). Individuals without a prior diagnosis had clinical OA confirmed by an orthopaedic surgeon or physiotherapist via telephone (diagnosis according to National Institute for Health and Care Excellence (NICE) criteria and Swedish National Guidelines, and confirming the absence of any red flag symptoms), or if deemed necessary were recommended to seek face-to-face care before inclusion in the programme.
* From October 1st 2021, all patients should have undergone a physical examination by doctor or physiotherapists before being able to enter the treatment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants with knee or hip OA that have joined the digital OA treatment program via online advertisements and campaigns placed on search engines and social networks, or by recommendations by their local physiotherapist or orthopaedic surgeon. Procedure for inclusion and exclusion has been described above.
  Data will be extracted from the Joint Academy (JA) database and the Better management of patients with OsteoArthritis (BOA) registry.
Sampling Method: Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Postal code/Official Municipality Key | Baseline
  Postal code/Official Municipality Key of participants
Postal code/Official Municipality Key for primary care center | Baseline
  For the BOA group only

CONTACTS AND LOCATIONS:
Overall Officials: Leif E Dahlberg, Senior professor, Study Director — Joint Academy
Locations (1):
- Joint Academy, Malmo, Sweden